CLINICAL TRIAL: NCT02170493
Title: Development and Clinical Trial of an Insole Sensor to Determine Optimal Limb Loading in the Rehabilitation of OTA Type 42IIIB and IIIC Lower Extremity Fractures
Brief Title: Insole Sensor to Determine Optimal Limb Loading
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: William Beaumont Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, David Rothberg, M.D., University of Utah
Other Study IDs: 58956
Record Dates: First submitted 2014-06-18; First posted 2014-06-23 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-08

CONDITIONS: Lower Extremity Fractures
Keywords: Insole Sensor; Optimial Limb Loading; 42IIIB; IIIC; Lower Extremity Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to use a novel load monitoring technology to correlate limb loading to OTA type 42IIIB and IIIC tibial fracture outcomes. This study will be the first to collect continuous limb loading data and will provide the first objective insight into how limb loading directs fracture healing. To meet this purpose, two specific aims have been developed.

Specific Aim 1: Preclinical validation of a load-monitoring insole

The Hitchcock laboratory has overcome the greatest technical hurdle for continuous limb load monitoring: development of load sensor technology that is affordable, accurate and capable of monitoring for over four weeks. To develop this sensor technology into a load-monitoring insole, the Hitchcock lab will incorporate consumer type electronics into the design, including a microprocessor, battery, and data storage media.

Following construction of a functional load-monitoring insole, a pilot human study with orthopaedic trauma patients from the University of Utah (N=20) will be conducted to identify modes of device failure, improve device interfacing and develop data handling protocols and software for the clinical arm of the proposed study.

Specific Aim 2: Conduct a prospective, direct observational cohort study.

Thirty (30) open tibial fracture patients will be recruited at two centers: University of Utah (N=15) and William Beaumont Army Medical Center (N=15). Participants will wear a walking boot instrumented with the load-monitoring insole that will continuously record limb loading and serve as a step counter. X-rays collected at standard-of-care follow-up visits will be used by Drs. Kubiak and Orr to subjectively evaluate fracture healing. A questionnaire regarding subjective perception of patient compliance will be collected at the first and last follow-up visits. Data collected from the insole sensor will be correlated to objective measures of fracture healing and subjective measures of patient compliance to determine the effect of patient limb loading on injury outcome. The Hitchcock laboratory will develop software to process and summarize data from the load monitoring insole and continually improve human interfacing factors of the load monitoring insole based off of feedback from the clinical team and study participants.

ELIGIBILITY:
Inclusion Criteria:

Specific Aim 1 Inclusion Criteria

* Patient is 18 years of age or older
* Patient has below the knee fracture
* Patient speaks English
* Patient weighs between 100 and 250 pounds
* Patient lives in close enough proximity to the the hospital to return for all appointments (~100 miles)

Specific Aim 2 Inclusion Criteria

* Patient is 18 years of age or older
* Patient has a tibia fracture
* Patient speaks English
* Patient weighs between 100 and 250 pounds
* Patient lives in close enough proximity to the the hospital to return for all appointments (~100 miles)

Exclusion Criteria:

Specific Aim 1 Exclusion Criteria

* Patient is younger than 18 years of age
* Patient does not have a below the knee fracture
* Patient does not speak English
* Patient weighs less than 100 pounds or more than 250 pounds
* Patient does not live in close enough proximity to the hospital to return for all appointments (~100 miles)
* Patient has another fracture that will alter his/her weight bearing status

Specific Aim 2 Exclusion Criteria

* Patient is younger than 18 years of age
* Patient does not have a tibia fracture
* Patient does not speak English
* Patient weighs less than 100 pounds or more than 250 pounds
* Patient does not live in close enough proximity to the hospital to return for all appointments (~100 miles)
* Patient has another fracture that will alter his/her weight bearing status

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who present to the University of Utah with an Open Tibial Fractures.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2013-01; Primary Completion 2017-07-10 (Actual); Study Completion 2017-07-10 (Actual)

PRIMARY OUTCOMES:
Patient Activity Measure (PAM-13) Questionnaire | Follow Up Visits up to 1-Year
  A subjective evaluation of perceived compliance with physician instruction

SECONDARY OUTCOMES:
X-ray (AP and Lateral) | Follow Up Visits up to 1 Year
  Subjectively evaluate fracture healing

CONTACTS AND LOCATIONS:
Overall Officials: David Rothberg, MD, Principal Investigator — Orthopedic Surgery
Locations (1):
- University of Utah, Salt Lake City, Utah, United States